CLINICAL TRIAL: NCT05912049
Title: A Phase 1, Randomized, Double-blind，Placebo-controlled, Single Ascending Dose Study to Evaluate the Safety, Tolerability, Pharmacokinetic, Pharmacodynamics and Immunogenicity of 9MW3811 in Healthy Participants
Brief Title: A Study to Evaluate the Safety, Tolerability, Pharmacokinetic Properties and Immunogenicity of 9MW3811 in Healthy Subjects
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Mabwell (Shanghai) Bioscience Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 9MW3811-2023-CP103
Record Dates: First submitted 2023-06-12; First posted 2023-06-22 (Actual); Last update posted 2023-09-01 (Actual); Status verified 2023-06

CONDITIONS: Idiopathic Pulmonary Fibrosis
MeSH Terms: conditions — Idiopathic Pulmonary Fibrosis

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 9MW3811 Injection (Experimental): single dose escalation for experimental drug
  Interventions: Drug: 9MW3811 Injection
- Placebo (Placebo Comparator): matching placebo administration for control
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: 9MW3811 Injection — Single dose intravenously infused on day 1
  Arms: 9MW3811 Injection
Drug: Placebo — Single dose of matching placebo intravenously infused on day 1
  Arms: Placebo

SUMMARY:
This is a single ascending dose study of 9MW3811, the primary objective of which is to evaluate the safety and tolerability of 9MW3811 in healthy adult participants.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female participants between 18 and 55 years of age, inclusive.
2. Male body weight ≥50.0 kg, or female body weight ≥45.0 kg, and body mass index (BMI) between 18.0 and 26.0 kg/m2, inclusive.
3. In good health determined by the investigator based on a medical evaluation.

Exclusion Criteria:

1. Clinically significant histories determined by the investigator of cardiovascular, hepatic, renal, gastrointestinal, neurological, respiratory, hematological, endocrinological, immunological, metabolic, and musculoskeletal abnormalities.
2. Having any history of an allergy to biological agents or any components of study drug; those who have a history of allergies and judged by the investigator to be ineligible for enrolment.
3. Use of any prescription medication 14 days prior to dosing or over-the-counter medication, vitamins, and/or herbal medicines 7 days prior to dosing (Excluding oral contraception, occasional paracetamol, ibuprofen and standard dose of multivitamins at the discretion of the PI or designee)
4. Participants who have been vaccinated within 4 weeks prior to screening or who are scheduled to be vaccinated during the study
5. Participants who received immunosuppressants except for previous use of inhaled or nasal corticosteroids 4 weeks earlier before administration or any oral corticosteroids 8 weeks earlier before administration, and who had received a single dose of monoclonal antibodies for any reason within 1 year prior to screening
6. Participants with one or more clinically significant positive test results of hepatitis B surface antigen (HBsAg), hepatitis C virus (HCV) antibody, treponema pallidum antibody or human immunodeficiency virus (HIV) antibody
7. History of active tuberculosis, or participants with active or latent tuberculosis infection during screening
8. History of drug abuse including narcotic and psychiatric drugs within 6 months prior to screening or a positive drug abuse test result at baseline (Morphine, Methamphetamine, Tetrahydrocannabinol acid)

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Estimated)
Dates: Start 2023-07-26 (Actual); Primary Completion 2023-12 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Incidence of adverse events (AEs) as assessed by CTCAE v5.0 | up to Day113
  An AE is any untoward medical occurrence in a patient or clinical investigation subject administered a pharmaceutical product and which does not necessarily have a causal relationship with this treatment.

SECONDARY OUTCOMES:
Maximum Plasma Concentration (Cmax) | up to Day113
  To determine the pharmacokinetic (PK) of 9MW3811 following single ascending intravenous doses in healthy adult participants.
Time to reach Cmax (Tmax) | up to Day113
  To determine the PK of 9MW3811 following single ascending intravenous doses in healthy adult participants.
Area under the plasma concentration versus time curve (AUC) from time 0 to the last quantifiable concentration (AUC0-t) | up to Day113
  To determine the PK of 9MW3811 following single ascending intravenous doses in healthy adult participants.
Terminal elimination half-life (t1/2) | up to Day113
  To determine the PK of 9MW3811 following single ascending intravenous doses in healthy adult participants.
AUC from time 0 extrapolated to infinity (AUC0-inf) | up to Day113
  To determine the PK of 9MW3811 following single ascending intravenous doses in healthy adult participants.
Terminal elimination rate constant (λz) | up to Day113
  To determine the PK of 9MW3811 following single ascending intravenous doses in healthy adult participants.
Apparent clearance (CL) | up to Day113
  To determine the PK of 9MW3811 following single ascending intravenous doses in healthy adult participants.
Volume of distribution (Vz) | up to Day113
  To determine the PK of 9MW3811 following single ascending intravenous doses in healthy adult participants.
Incidence of antidrug antibodies (ADA) at specified timepoints relative to baseline | up to Day113
  To determine the immunogenicity of 9MW3811.

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital of Soochow University, Suzhou, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No